## INFORMED CONSENT FORM

in relation to the research project: "Fostering Ukraine's capacity in delivery and research of innovative evidence-based PTSD treatment (Lux4UA)"

| I, | , have read and understood the information |
|---|---|
| sheet regarding the above-mentioned research project | (Lux4UA Project) conducted by the research |
| team from the University of Luxembourg (UNILU), th | e Centre of Mental Health and Rehabilitation |
| "Forest Glade" of the Ministry of Health of Ukraine (R | CFG), the National Psychological Association |
| of Ukraine (NPAU). I have been informed orally and i | n writing about the nature, purpose, duration, |
| procedures, potential risks, and benefits of participatin | g in the Lux4UA Project, and I have had the |
| opportunity to ask questions. | |

I understand that the Lux4UA Project aims to evaluate the effectiveness and feasibility of the Reconsolidation of Traumatic Memories (RTM) Protocol for PTSD treatment in Ukraine. My participation involves training in the RTM Protocol, delivering the RTM Protocol and treatment-asusual (TAU) to assigned clients, collecting clients' data, and participating in the feasibility study through surveys and focus group interviews.

## I understand that:

- Participation is voluntary.
- My personal data will be processed according to the EU General Data Protection Regulation (GDPR) and the Law of Ukraine on the Protection of Personal Data.
- My personal data (name, contact details, education, workplace, etc.) and opinions of the RTM Protocol will be collected and stored securely on protected servers in Ukraine for training, certification, and study coordination and will not be transferred to Luxembourg.
- Data used for research purposes will be anonymised.
- I may contact the research team at any time to object to further processing or request deletion of my personal data.

## Please indicate your consent below:

| Statement | Yes | No |
|---|---|---|
| I consent to the collection and processing of my personal data for participation in the professional training and research activities. | | |
| I agree to participate in surveys and focus group interviews to evaluate the feasibility of the RTM Protocol. | | |
| I consent to my survey answers being used for the purposes of the Research Project in anonymized form. | | |
| I consent to my interviews (from participation in focus-group interview) being recorded in audio format and being used for the purposes of the Research Project in anonymized form. | | |
| I agree to the data I provide being archived and used in anonymised form for other research in the metal health area beyond the Lux4UA Project. | | |
| I consent to my responses being used in anonymised form for research publications and policy recommendations. | | |

| I consent to being contacted for possible participation in a follow-up study or future collaboration. | |
|---|---|
| I voluntarily agree to take part in the Lux4UA Project. | |
| PARTICIPANT | |
| Last name: | |
| First name: | |
| Email-address | |
| Phone number | |
| Place & date: | |
| Signature: | |
| RESEARCH COORDINATOR I have explained the purpose, procedures, risks, and benefits of the Lux4UA Project to participant named above and answered all their questions. Last name: | the |
| First name: | |
| Place & date: | |
| Signature: | |
| Data-related contacts: | |

NPA Data Protection Officer (email: <a href="mailto:dpo@npa-ua.org">dpo@npa-ua.org</a>; address: 12 Kozhumiatska Street, 04071, Kyiv, Ukraine (Nadia Diatel)

RCFG Protection Officer (email: dataprotection.forestglade@mailbox.org; address: 25, Line 7, Puscha-Vodytsia, 04114, Kyiv, Ukraine (Marta Vulchyn)